CLINICAL TRIAL: NCT00335218
Title: A Multi-center, Prospective, Randomized, Double-blind, Placebo-controlled, Two-arm, Phase IV Study to Investigate the Influence of a Continuous Combined Estrogen-progestin Regimen Containing 2 mg Estradiol Valerate and 2 mg Dienogest (Climodien® / Lafamme®) on the Fat Distribution in Otherwise Healthy Early Postmenopausal Women
Brief Title: Fat Distribution in Healthy Early Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91161; 306387
Record Dates: First submitted 2006-02-24; First posted 2006-06-09 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Healthy; Postmenopause
Keywords: Early postmenopausal state; Climacteric symptoms; Hormone replacement therapy
MeSH Terms: interventions — estradiol valerate-dienogest

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Climodien / Lafamme (BAY86-5027)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Climodien / Lafamme (BAY86-5027) — 1 tablet daily (2 mg EV + 2 mg DNG)
  Arms: Arm 1
Drug: Placebo — 1 tablet daily
  Arms: Arm 2

SUMMARY:
The aim of this study is to explore the effects of hormone replacement therapy with EV/DNG on abdominal fat distribution measured by magnetic resonance imaging.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy early postmenopausal women
* BMI between 25 and 30

Exclusion Criteria:

* Contra-indication(s) for hormone treatment
* Metabolic diseases
* Concomitant medication with influence on lipid metabolism

Ages: 48 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2002-07; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Individual relative change of abdominal visceral fat measured by magnetic resonance imaging | Baseline and after 24 weeks of treatment

SECONDARY OUTCOMES:
Parameters of body composition and lipid metabolism | Baseline and after 24 weeks of treatment
Adverse events collection | During whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Austria (2):
  - Vienna, Vienna
  - Vienna